CLINICAL TRIAL: NCT00602160
Title: Investigation of the Efficacy of the Food Allergy Herbal Formula (FAHF-2TM) in Patients With Food Allergy - Phase II Trial
Brief Title: Therapeutic Effect of Chinese Herbal Medicine on Food Allergy
Acronym: FAHF-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li, Xiu-Min, M.D. (Individual)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Xiu-Min Li, M.D., Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: R01AT001495-01A1 (NIH); R01AT001495-01A1 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Food Allergy
Keywords: Food allergy; Chinese Herbs; Investigational new drug; Herbs; Therapeutic medicine; Traditional Chinese medicine
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 2 different dosages
  Interventions: Drug: FAHF-2 (TM)
- 2 (Placebo Comparator)
  Interventions: Drug: FAHF-2 (TM)

INTERVENTIONS:
Drug: FAHF-2 (TM) — We propose to test 10 tablets administered orally three times daily (t.i.d.) for 6 months in the Phase II study. The subjects will be randomized to 1 of 2 groups; FAHF-2 or Placebo group.
  Both groups will undergo physician supervised Double-blinded placebo controlled food challenges, once during screening before starting treatment and again after 6 months of therapy.

SUMMARY:
The increasing prevalence of allergic diseases in westernized countries poses a significant health problem and a tremendous burden on quality of life and healthcare expenditure. Food allergy affects as many as 6% of young children and 3% to 4% of adults. While the majority of children outgrow their allergy to milk, egg, wheat and soy, allergies to peanut, tree nuts, fish and shellfish are often life-long. Currently, there are no treatments that can cure or provide long-term remission from food allergy. Based on our preliminary studies, we hypothesize that our investigational botanical drug, FAHF-2TM, will be a safe and effective herbal therapy for food allergy. We are enrolling those age 12-45 yrs old with allergies to peanut, tree nuts, sesame, fish, and/or shellfish.

DETAILED DESCRIPTION:
To address our hypothesis, we propose the following aims:

Aim #1: To investigate the efficacy of FAHF-2TM for food allergy (in addition to current food allergen avoidance).

Aim #2: To characterize the immunomodulatory effects of FAHF-2TM on food allergic patients

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 12 through 45 years of age and otherwise in good health as determined by medical history and physical examination
* History of allergy to peanut, tree nut, sesame, fish or shellfish as documented by a positive skin test and/or food allergen-specific IgE level.
* The subject agrees to participate in the study or the subject's parent or legal guardian is willing and able to give written informed consent, and the pediatric subject gives assent for participation in the study.
* Positive double-blind placebo controlled food challenge to peanut, tree nuts, sesame, fish, or shellfish.
* Females of childbearing potential must be inactive sexually or take effective birth control measures, as deemed appropriate by the investigator, for the duration of the study

Exclusion Criteria:

* History of life-threatening anaphylaxis to peanut, tree nut, sesame, fish or shellfish (involving hypotension or requiring mechanical ventilation)
* Allergy to corn
* Acute febrile illness (such as cold, flu, etc.) within one week before administration of study drug
* Any history of systemic disease that in the investigator's opinion would preclude the subject from participating in this study, e.g. autoimmune disease, neoplasms, HIV or hepatitis virus infection
* Allergic gastrointestinal disease (e.g. allergic eosinophilic esophagitis/gastroenteritis
* Abnormal hepatic function (ALT/AST and bilirubin >1.25 x upper limit of normal)
* Abnormal bone marrow function (WBC <4 x 103/mm3; platelets <100 x 103/mm3; hgb <11 g/dl)
* Abnormal renal function (BUN and creatinine >1.25 x upper limit of normal)
* Clinically significant abnormal electrocardiogram
* Current uncontrolled moderate to severe asthma as defined by:

  1. FEV1 value <80% predicted or any clinical features of moderate or severe persistent asthma baseline severity (as defined by the 2007 NHLBI Guidelines) and greater than high daily doses of inhaled corticosteroids (as defined for children and adults using dosing tables from the 2007 NHLBI Guidelines).
  2. Use of steroid medications in the following manners: history of daily oral steroid dosing for >1 month during the past year, or burst or steroid course in the past 6 months, or >1 burst oral steroid course in the past year.
  3. Asthma requiring >1 hospitalization in the past year for asthma or >1 ED visit in the past 6 months for asthma.
* Participation in another experimental therapy study within 30 days of this study
* History of alcohol or drug abuse
* Currently taking antidepressant medication
* Pregnant or lactating female subjects. Females of childbearing potential will need a negative serum pregnancy test at screening to be considered for this study
* Use of omalizumab
* Use of beta blockers, ACE inhibitors, ARB, or calcium channel blockers, or history of ischemic heart disease
* Inability to discontinue use of antihistamines for skin testing or oral food challenges
* Inability to take the tablets

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety of FAHF-2 | 1 year

SECONDARY OUTCOMES:
lab studies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wang, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Xiu-Min Li, Study Director — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mount Sinai School Medicine, New York, New York

REFERENCES:
- [Derived] Wang Z, Wang ZZ, Geliebter J, Tiwari R, Li XM. Traditional Chinese medicine for food allergy and eczema. Ann Allergy Asthma Immunol. 2021 Jun;126(6):639-654. doi: 10.1016/j.anai.2020.12.002. Epub 2020 Dec 10. PMID 33310179
- [Derived] Wang J, Jones SM, Pongracic JA, Song Y, Yang N, Sicherer SH, Makhija MM, Robison RG, Moshier E, Godbold J, Sampson HA, Li XM. Safety, clinical, and immunologic efficacy of a Chinese herbal medicine (Food Allergy Herbal Formula-2) for food allergy. J Allergy Clin Immunol. 2015 Oct;136(4):962-970.e1. doi: 10.1016/j.jaci.2015.04.029. Epub 2015 Jun 1. PMID 26044855
- [Derived] Song Y, Wang J, Leung N, Wang LX, Lisann L, Sicherer SH, Scurlock AM, Pesek R, Perry TT, Jones SM, Li XM. Correlations between basophil activation, allergen-specific IgE with outcome and severity of oral food challenges. Ann Allergy Asthma Immunol. 2015 Apr;114(4):319-26. doi: 10.1016/j.anai.2015.01.006. PMID 25841330
- [Derived] Noone S, Ross J, Sampson HA, Wang J. Epinephrine use in positive oral food challenges performed as a screening test for food allergy therapy trials. J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):424-8. doi: 10.1016/j.jaip.2014.10.008. Epub 2015 Jan 13. PMID 25609353
- [Derived] Yang N, Wang J, Liu C, Song Y, Zhang S, Zi J, Zhan J, Masilamani M, Cox A, Nowak-Wegrzyn A, Sampson H, Li XM. Berberine and limonin suppress IgE production by human B cells and peripheral blood mononuclear cells from food-allergic patients. Ann Allergy Asthma Immunol. 2014 Nov;113(5):556-564.e4. doi: 10.1016/j.anai.2014.07.021. Epub 2014 Aug 22. PMID 25155085
- [Derived] Patil SP, Wang J, Song Y, Noone S, Yang N, Wallenstein S, Sampson HA, Li XM. Clinical safety of Food Allergy Herbal Formula-2 (FAHF-2) and inhibitory effect on basophils from patients with food allergy: Extended phase I study. J Allergy Clin Immunol. 2011 Dec;128(6):1259-1265.e2. doi: 10.1016/j.jaci.2011.06.015. Epub 2011 Jul 26. PMID 21794906
- [Derived] Wang J, Patil SP, Yang N, Ko J, Lee J, Noone S, Sampson HA, Li XM. Safety, tolerability, and immunologic effects of a food allergy herbal formula in food allergic individuals: a randomized, double-blinded, placebo-controlled, dose escalation, phase 1 study. Ann Allergy Asthma Immunol. 2010 Jul;105(1):75-84. doi: 10.1016/j.anai.2010.05.005. PMID 20642207